CLINICAL TRIAL: NCT05327049
Title: Evaluation of the Remineralizing Effect of Aloe Vera Versus Diode Laser for Management of Deep Carious Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hayam mosad, Assistant lecturer of operative dentistry, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPEN- 108-L
Record Dates: First submitted 2022-04-06; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Deep Caries
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no intervention (Experimental): No Intervention: conventional selective caries removal without treatment After taking the first sample of dentin, the cavity will be restored
  Interventions: Other: no intervention
- diode laser treatment (Experimental): After selective caries removal the cavity was irradiated in contact mode with continuous wave of radiation through a 400µm flexible fiber that was inserted inside the cavity with a spiral continuous movement clockwise from the top to the floor and anti-clockwise in the reverse direction. Irradiation time was 15 seconds and repeated three times for 15 seconds interval with contact, pulsed mode and the output power was adjusted at 1.30 Watt.
  Interventions: Device: diode laser
- Aloe Vera treatment (Experimental): After selective caries removal the lesions were treated with aloe Vera paste which was prepared by mixing aloe Vera powder by distilled water until a thick paste is formed. the paste was applied to the prepared floor by condenser to cover the remaining carious lesion
  Interventions: Dietary Supplement: Aloe Vera

INTERVENTIONS:
Other: no intervention — treatment of deep carious lesions
  Arms: no intervention
Device: diode laser — laser light for cavity disinfection
  Arms: diode laser treatment
Dietary Supplement: Aloe Vera — herbal dietary supplement for treatment of deep carious lesions
  Arms: Aloe Vera treatment

SUMMARY:
The present study will be performed to evaluate:

The remineralizing effect of Aloe Vera versus Diode laser on deep carious dentin after selective caries removal.

DETAILED DESCRIPTION:
This study was conducted on 45 teeth selected from patients according to inclusion and exclusion criteria. They were selected from the dental clinic in faculty of oral and dental medicine for girls, Al-Azhar University. The procedure was explained and written informed consent was obtained from each patient. The possible discomforts, risks, and benefits were fully explained to the patients. Ethical committee approval was obtained.

Protocol of caries removal was Applied Subsequently, the central cariogenic biomasses and superficial part of the necrotic and demineralized dentin was excavated, leaving the leathery dentin layer.

Sample grouping:

The patients were randomly assigned into three main groups according to the material used (15 for each) which were assessed at different time intervals (B1) after three months,(B2) after six months.

A1: cavities will be sealed directly by temporary restorative material (conventional glass ionomer) without any treatment.

A2: cavities will be treated by Diode laser then sealed directly by temporary conventional glass ionomer.

A3: cavities will be treated with Aloe Vera then sealed directly by temporary conventional glass ionomer.

Evaluation of the remineralization effect of Each group will be assessed radiographically immediately at base line (B0), after three months (B1) and six months (B2) to evaluate the dentin remineralization.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have active deep carious lesion.
* clinical and radiographic examinations of carious lesions.

Exclusion Criteria:

* Teeth with pulpal involvement
* Teeth with abscess
* Teeth with pain or swelling
* Teeth with developmental disorders
* Teeth with adjacent soft tissue lesions
* patients with systemic illness will be excluded

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
assessment of the remineralizing effect of aloe vera and diode laser on deep caries | 6 months
  remineralisation will be assessed by radiodensity using digital radiography

CONTACTS AND LOCATIONS:
Overall Officials: Maha Niazy, professor, Study Director — Al-Azhar University
Locations (1):
- Al-Azhar University, Naşr, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No